CLINICAL TRIAL: NCT00380601
Title: An Open-label, PhaseⅢ Study to Evaluate the Efficacy and Safety of MRA in Patients With RA
Brief Title: PhaseⅢOpen-label Study of MRA for Rheumatoid Arthritis(RA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Chugai Pharmaceutical Co.,Ltd., Chugai Pharmaceutical Co.,Ltd.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRA225JP
Record Dates: First submitted 2006-09-25; First posted 2006-09-26 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: MRA(Tocilizumab)

INTERVENTIONS:
Drug: MRA(Tocilizumab) — 8mg/kg/4 weeks

SUMMARY:
An open-label, PhaseⅢ study to evaluate the efficacy and safety of MRA in patients with RA

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as having RA, on the basis of the criteria stipulated by the American Conference on Rheumatism(ACR) in 1987
* Active RA despite at least one DMARDs or immunosuppressants or Infliximab or Etanercept.Active disease is defined as having at least 6 tender and 6 swollen joints among DAS28 (Modified Disease Activity Scores that include twenty eight joint counts) and ESR at least 30 mm/hr or CRP not less than 2.0mg/dL
* Active RA despite over 10mg adrenocortical steroids within 2 weeks before entry of this study

Exclusion Criteria:

* Shown to have class-Ⅳ Steinbrocker's functional activity in an evaluation carried out within 4 weeks before administration of the study drug
* Treated with Infliximab within 3 months before and with Etanercept within 2 weeks before administration of the study drug
* Subjected to any of the following within 4 weeks before administration of the study drug:

  1. Surgical treatment (operations,etc.).
  2. Plasma exchange method

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-05; Primary Completion 2008-08 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Frequency of ACR 20％ improvement at the final visit | throughout study

SECONDARY OUTCOMES:
Time course of the frequency of ACR 20％, 50％ and 70％ improvement,time course of individual items within the ACR core set. | throughout study
Time course of DAS28 to the final visit. | throughout study
Time course of steroid sparing effect from first visit to final visit. | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Yuji Kimura, Study Director — Chugai Pharmaceutical Co., Ltd. Research Dept.1
Locations (10):
- Japan (10):
  - Chugoku region, Chugoku
  - Chukyo region, Chukyo
  - Hokkaido region, Hokkaido
  - Hokuriku region, Hokuriku
  - Kansai region, Kansai
  - Kanto region, Kanto
  - Kousinetsu region, Kousinetsu
  - Kyushu region, Kyushu
  - Sikoku region, Sikoku
  - Tohoku region, Tōhoku